CLINICAL TRIAL: NCT06475521
Title: A Randomised, Controlled, Double-blinded, Multi-country, Multi-centre Trial to Study Growth and Health Outcomes of a New Infant- and Follow-on Formula for Healthy Term Infants.
Acronym: GAIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SBB22R&56319
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-06

CONDITIONS: Baby Formula, Growth Equivalence, Neurocognitive Development, Healthy Infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, double-blinded, multi-country, multi-center
  Including Breastfed reference group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Infant formula test group; Group that receives the test product.
  Interventions: Other: Infant Formula
- Arm 2 (Active Comparator): Infant formula control group; Group that receives a comparative control product.
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula — Test group

SUMMARY:
To demonstrate growth equivalence of a Baby formula Test Product when compared to the Control product after 16 weeks. And to demonstrate better neurocognitive development at 52 weeks post-baseline in subjects receiving the Test Product, compared to subjects receiving the Control Product. Also, other anthropometric parameters will be investigated up to 52 weeks.

A Breastfed reference group, exclusively breastfed for at least 16 weeks, will also be included.

DETAILED DESCRIPTION:
The study will include infants to be randomised to receive the Test or Control product for 52, and infants whose parents have the intention to provide exclusively breastfeeding for at least 16 weeks after enrolment. Baseline assessments will be done at Visit 1/enrolment visits.

Subjects will return for clinic visits at 2 (Visit 2), 4 (Visit 3), 8 (Visit 4), 12 (Visit 5), 16 (Visit 6) 26 (Visit 7), 39 (Visit 8), and 52 (Visit 9) weeks post-baseline. During these clinic visits the investigator will perform anthropometric measurements, interview parent(s) about their infant's product intake/breastfeeding, occurrence of (serious) adverse events, medication/nutritional supplement use, details of infections and antibiotic/antiviral usage (if applicable).

At selected visits the following will be assessed a) stool characteristics (V2, 4, 6, 7,8, 9)); b) type of weaning food introduction (as of V6); c) neurocognitive development (V9); d) a three-day 24 hour food recall for dietary intake; e) stool samples at (V1, 6, 9); and f) blood sample (V6).

Also, a follow-up phone call is planned 2 weeks after the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton, term born infants (gestational age ≥ 37 weeks + 0 days and ≤ 41 weeks + 6 days).
* Infants aged ≤ 14 days at enrolment.
* Weight at birth within 10th to 90th percentile per gestational age and sex, according to Intergrowth Standards
* For formula feeding groups: Infants fully formula fed at the time of enrolment.
* For breastfed reference group: Infants exclusively breastfed at the time of enrolment and parent(s) intend to exclusively breastfeed the infant at least until 16 weeks after Visit 1.
* Written informed consent (IC) from parent(s) and/or legally acceptable representative(s) aged ≥18 years at enrolment.

Exclusion Criteria:

* . Infants who require a special diet other than IF with intact cow's milk protein.
* Infants known or suspected to have cow's milk, fish, and/or soy allergy and/or lactose intolerance.
* Infants with current or previous illnesses/conditions and/or known or suspected congenital diseases or malformations which could interfere with the study outcomes, as per investigator's clinical judgement.
* Infants whose mother is known to suffer from an illness or condition which could interfere with the study outcomes, as per investigator's clinical judgement.
* Infants with previous, current, or intended participation in any concomitant clinical study involving investigational or marketed products.
* Investigator's uncertainty about the willingness or ability of parents or legally acceptable representative(s) to comply with the protocol requirements.

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 579 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight gain | Baseline to 16 weeks post-baseline
  To demonstrate equivalence in mean weight gain per day from baseline to 16 weeks post-baseline in subjects receiving the Test product, compared to subjects receiving the Control product

SECONDARY OUTCOMES:
Neurocognitive Development | 52 weeks post baseline
  Demonstrate better neurocognitive development as measured by the Bayley Scales of Infant and Toddler Development (Bayley-3) cognitive composite score at 52 weeks post-baseline in subjects receiving the Test product, compared to subjects receiving the Control product.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Asklepiy OOD Dupinista, Dupnitsa, Bulgaria

IPD SHARING:
Plan to Share IPD: No